CLINICAL TRIAL: NCT02691351
Title: Intercontinental Cooperative Non-Hodgkin T-cell Lymphoma Prospective Registry Study
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Principal Investigator, Samsung Medical Center
Other Study IDs: 2015-11-070
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Non-Hodgkin T-cell Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- non-Hodgkin T-cell Lymphoma
  Interventions: Other: Prospective Registry

INTERVENTIONS:
Other: Prospective Registry — Survival and disease status follow-up at 1st primary treatment, 1st salvage treatment and 2nd salvage treatment
  1. Regimen
  2. Response Evaluation
  3. SUSAR(Suspected, Unexpected, Serious, Adverse Reaction) collection

SUMMARY:
The better understanding of non-Hodgkin T-cell lymphoma is essential for establishing effective treatment strategy for non-Hodgkin T-cell lymphoma. Therefore, the data about conical features and treatment outcomes of each subtype should be accumulated to establish treatment strategy. However, the majority of previous data for non-Hodgkin T-cell lymphoma was from small case series of single institute. Furthermore, as novel drugs were developed for the treatment of relapsed or refractory T-cell lymphoma, the date from patients who were treated with those novel drugs are especially required because their outcomes may reflect the outcomes of currently available treatments. Thus, a multinational, multicenter prospective registry study is needed to provide information useful for establishing treatment strategies for T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed Mature T-cell non-Hodgkin lymphoma based on the World Health Organization classification 2008
* Newly diagnosed patients without a previous treatment history for T-cell lymphoma or relapsed/refractory T-cell lymphoma patients
* Age ≥19 years
* Written informed consent

Exclusion Criteria:

* Hodgkin lymphoma
* non-Hodgkin B-cell lymphoma
* Immature non-Hodgkin T-cell lymphoma: Precursor T-lymphoblastic lymphoma/leukemia
* Not understanding informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T-cell non-Hodgkin lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Overall response rate to primary treatment and salvage treatment | 5 years
Progression-free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Won seog Kim, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea